CLINICAL TRIAL: NCT05970744
Title: Randomized, Double-blind, Placebo-controlled Phase 1 Trial of the RSV/Flu-01E Vaccine for the Prevention of Respiratory Syncytial Virus Infection in Volunteers Aged 18 to 59 Years and Over 60 Years
Brief Title: Evaluation of RSV/Flu-01E Vaccine for the Prevention of RSV Infection in Volunteers Aged 18 to 59 Years and Over 60 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tatyana Zubkova (Other)
Responsible Party: Sponsor-Investigator, Tatyana Zubkova, Head of the clinical department, Research Institute of Influenza, Russia
Organization: Research Institute of Influenza, Russia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RSV-I-01/2022; 736 30.12.2022 (Other: Russian Clinical Trial Authorization Registry [RCT])
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus infection; Vaccine; Influenza vector; Intranasal immunization
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- RSV/Flu-01E low dose 18-59 (Experimental): Participants aged 18 to 59 years will receive single injection of low dose RSV/Flu-01E Vaccine
  Interventions: Biological: RSV/Flu-01E low dose
- RSV/Flu-01E high dose 18-59 (Experimental): Participants aged 18 to 59 years will receive single injection of high dose RSV/Flu-01E Vaccine
  Interventions: Biological: RSV/Flu-01E high dose
- Placebo 18-59 (Placebo Comparator): Participants aged 18 to 59 years will receive single injection of Placebo
  Interventions: Biological: Placebo
- RSV/Flu-01E high dose over 60 (Experimental): Participants aged over 60 years will receive single injection of high dose RSV/Flu-01E Vaccine
  Interventions: Biological: RSV/Flu-01E high dose
- Placebo over 60 (Placebo Comparator): Participants aged over 60 years will receive single injection of Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV/Flu-01E low dose — Participants will receive single intranasal injection of A/H1N1pdm09 recombinant attenuated influenza vector (7.7 lg EID50) with modified NS gene coding for the F antigen of respiratory syncytial virus
  Arms: RSV/Flu-01E low dose 18-59
Biological: RSV/Flu-01E high dose — Participants will receive single intranasal injection of A/H1N1pdm09 recombinant attenuated influenza vector (8.4 lg EID50) with modified NS gene coding for the F antigen of respiratory syncytial virus
  Arms: RSV/Flu-01E high dose 18-59; RSV/Flu-01E high dose over 60
Biological: Placebo — Participants will receive single intranasal injection of Placebo
  Arms: Placebo 18-59; Placebo over 60

SUMMARY:
The aim of the study is to investigate the safety and immunogenicity of the RSV/Flu-01E vaccine for the prevention of respiratory syncytial virus infection in volunteers aged18 to 59 years and over 60 years.

DETAILED DESCRIPTION:
Study includes 60 participants in three cohorts. First cohort includes 15 volunteers aged 18 to 59, randomized at 2:1 ratio, to receive low dose RSV/Flu-01E vaccine or placebo, correspondingly. Second cohort includes 15 volunteers aged 18 to 59, randomized at 2:1 ratio, to receive high dose RSV/Flu-01E vaccine or placebo, correspondingly. Third cohort includes 30 participants aged 60 years and older, randomized at 2:1 ratio to receive high dose RSV/Flu-01E vaccine or placebo. Duration of the study for each participant is about 6 months (no more than 190 days).

ELIGIBILITY:
Inclusion Criteria:

For the first and second cohort:

1. Availability of signed informed consent.
2. Adult men and women aged 18-59 years.
3. Diagnosed "healthy", according to the data of standard clinical, laboratory and instrumental examination methods provided for in this protocol, with the absence of clinically significant changes.
4. BMI from 18 to 30 kg/m2.
5. Individuals with antibody titer to influenza A/H1N1pdm09 ≤1:20 according to HI assay.
6. Ability and willingness to independently keep records in the diary of self-observation and carry out all visits according to the protocol.
7. Negative urine test for psychotropic and narcotic substances.
8. Negative breath alcohol test.
9. Consent of study participants to use effective contraceptive methods throughout their participation in the study. In this study, volunteers can use the following methods of contraception:

   * Combined methods:

     * male condom and spermicide
     * cervical cap and spermicide
     * vaginal diaphragm and spermicide
   * Intrauterine device
   * Hormonal intrauterine device
   * Hormonal contraceptives:

     * hormonal implants
     * hormone injections
     * combined oral contraceptives
     * mini-pill
     * contraceptive patch
   * Abstinence from sexual activity.
10. For women of childbearing potential - a negative pregnancy test.
11. Indicators of general and biochemical blood tests at screening within 1.1 x the upper limit - 0.9 x the lower limit of the reference intervals.
12. Negative tests for HIV, hepatitis B and C, syphilis.

For the third cohort:

1. Availability of signed informed consent.
2. Adult men and women over the age of 60.
3. The diagnosis is "healthy", verified according to standard clinical, laboratory and instrumental methods of examination or the presence of a chronic disease, if the researcher considers it to be compensated.
4. BMI from 18 to 30 kg/m2.
5. Individuals with antibody titer to influenza A/H1N1pdm09 ≤1:20 according to HI assay.
6. The ability and readiness to independently keep records in the diary of self-observation and carry out all the visits provided for in the study, provided for by the protocol.
7. Negative urine test for psychotropic and narcotic substances.
8. Negative breath alcohol test.
9. Indicators of general and biochemical blood tests for screening within 1.1 x the upper limit - 0.9 x the lower limit of the reference intervals.
10. Negative tests for HIV, hepatitis B and C, syphilis.

Exclusion Criteria:

1. Participation in another clinical study within three months prior to the start of the current study; planning to participate in another study during the current study period.
2. Contact with COVID-19 patients within 14 days prior to the start of the clinical study.
3. Positive rapid test result for SARS-CoV-2 antigen.
4. Immunization with any other non-study vaccine product within three weeks prior to enrollment in the current study, or refusal to postpone such until the end of the three-week period after completion of the current study.
5. Regular use of nasal irrigation therapy during the last six months prior to enrollment in the current study or episodic use of the above method of treatment in the two weeks prior to the screening.
6. History of frequent nosebleeds (>5) during the year prior to the current study
7. Anatomical features of the nose that may interfere with intranasal administration of the study drug
8. The presence of surgical intervention in the sinus area, paranasal sinuses, or traumatic injuries of the nose within a month before screening.
9. Symptoms of acute respiratory disease at the time of screening or within two weeks prior to screening.
10. Treatment with immunoglobulins or other blood derived medications in the three months prior to screening or planning such treatment during the period of participation in the current study.
11. Donation of blood/plasma (450 ml or more) less than 2 months prior to screening.
12. The presence or suspicion of the presence of various immunosuppressive or immunodeficiency conditions or continuous use (the drug was prescribed for more than 14 days without a break) of immunosuppressive drugs, immunomodulators for 6 months before the screening.
13. History of bronchial asthma.
14. Hypersensitivity and the presence of severe allergic reactions, including Quincke's edema, anaphylactic shock after the previous administration of any vaccine.
15. History of wheezing after previous immunization with live influenza vaccine.
16. Other adverse events after immunization (fever above 40°C, syncope, non-febrile convulsions, anaphylaxis) when there is a minimal likelihood that they are associated with a previous administration of any vaccine.
17. Suspicion of hypersensitivity to any component of the study vaccine, including egg protein.
18. Burdened allergic anamnesis.
19. Acute or chronic clinically significant lung, cardiovascular, hepatic, endocrine, neurological, or psychiatric disorders, or impaired renal function identified by history, physical examination, or clinical laboratory findings that, in the opinion of the investigator, may influence the outcome of the study.
20. History of oncological diseases.
21. History of thrombocytopenic purpura or bleeding disorders.
22. History of convulsions
23. Tuberculosis or residual changes after tuberculosis according to the anamnesis and / or available medical documentation.
24. Chronic alcohol dependence or chronic use of illicit drugs, drug abuse.
25. Claustrophobia and social phobia according to history and / or available medical records.
26. For women of reproductive age - lactation, pregnancy or suspected pregnancy, early postpartum period.
27. Inability to read in Russian; inability or unwillingness to understand the essence of the study. Any other condition that limits the eligibility of obtaining informed consent or may affect the volunteer's ability to participate in the study.
28. Military or law enforcement officers, persons serving sentences in places of deprivation of liberty or in custody.
29. Special diet (eg, vegetarian, vegan, salt-restricted) or lifestyle (night work, extreme physical activity)
30. Any condition that, in the opinion of the investigator, may increase the risk to the health of a volunteer participating in the study or affect the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with local and systemic adverse events (AEs) and serious adverse events (SAEs) | Throughout the study, average of 6 months
  * Adverse events (AEs) and serious AEs (SAEs), both vaccine related and non-vaccine related.
  * AEs/SAEs of particular importance:
    * Immediate AEs (allergic reactions) occurring within two hours of vaccination.
    * Post-vaccination reactions (anticipated clinical manifestations of a local and systemic nature), usually due to intranasal vaccination between two hours and the next 7 days after vaccination.
  * Evaluation of influenza A virus shedding evaluated by immunochromatographic rapid test in nasal swab samples in control points after vaccination

SECONDARY OUTCOMES:
Level of RSV F antigen-specific cytokine producing T-cells | Days 1, 7, 28, 90, 180
  Change from baseline in the level of cytokine producing CD4+ and CD8+ T-cells upon in vitro stimulation of PBMC with RSV F-peptide epitopes measured by ICS/ELISPOT
Level of RSV F antigen-specific cytokine release in whole blood assay | Days 1, 7, 28
  Change from baseline in the cytokine concentration in whole-blood cytokine release assay upon in vitro stimulation with RSV F-peptide epitopes measured in ELISA
Level of RSV F antigen-specific mucosal IgA antibody in saliva/nasal secrets | Days 1, 28
  Change from baseline in the level of secretory IgA antibody specific to RSV F-antigen measured in ELISA in nasal secret/saliva
Level of RSV F antigen-specific IgG antibody | Days 1, 28, 90, 180
  Changes in the levels of RSV F antigen-specific total serum IgG antibodies measured in ELISA in serum
Proportion of responders to vaccination | Days 7, 28
  Proportion of participants who responded to vaccination by significant increase in any of the immunogenicity parameters at any of the time points. The increase is considered significant if the fold change of the parameter value exceeds the conventional threshold, measured as geometric mean fold change in Placebo group multiplied by two geometric mean standard deviations.
Concentration of cytokines in nasal secrets after vaccination | Days 1, 2, 3
  Change from baseline in the concentration of cytokines in nasal secrets measured in ELISA (pg/ml, 13-plex assay, IFN-α2, TSLP, IL-1α, IL-1β, GM-CSF, IL-11, IL-12p40, IL-12p70, IL-15, IL-18, IL-23, IL-27, IL-33)
Influenza specific systemic antibody immune response | Days 1, 28
  Change from baseline in the titer of influenza specific antibodies in serum measured in hemagglutination inhibition/microneutralization assay
Influenza specific local antibody immune response | Days 1, 28
  Change from baseline in the level of influenza specific IgA antibodies in nasal secret/saliva measured in ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Zubkova, PhD, Principal Investigator — Smorodintsev Research Institute of Influenza
Locations (1):
- Smorodintsev Research Institute of Influenza, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No